CLINICAL TRIAL: NCT07301437
Title: A Real-world Study of Liraglutide Alone and in Combination With Orlistat for Weight Loss in Overweight/Obese Patients.
Brief Title: RWS of of Liraglutide Alone and in Combination With Orlistat for Weight Loss in Overweight/Obese Patients.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2025-202
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Overweight and Obese Adults
MeSH Terms: conditions — Overweight | interventions — Orlistat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Drug: liraglutide combined with orlistat
- control group (Active Comparator)
  Interventions: Drug: liraglutide monotherapy

INTERVENTIONS:
Drug: liraglutide monotherapy — liraglutide monotherapy
  Arms: control group
Drug: liraglutide combined with orlistat — combination therapy
  Arms: experimental group

SUMMARY:
To evaluate the differences in weight loss between liraglutide monotherapy and combined with orlistat in overweight/obese patients.

ELIGIBILITY:
Inclusion Criteria:

- 1.BMI: ≤ 35 kg/m² and ≥ 30 kg/m², or ≥ 27 kg/m² and having at least one obesity-related complication (such as hypertension, type 2 diabetes, dyslipidemia) 2.Voluntarily sign the informed consent form, agreeing to cooperate in completing the 24-week treatment and follow-up.

3.No severe cognitive impairment or mental illness, and able to understand and comply with the research requirements.

Exclusion Criteria:

* 1. Allergy to liraglutide, orlistat or excipients 2.Severe liver and kidney dysfunction: ALT or AST> three times the upper limit of normal, or eGFR <30 mL/min 3.Thyroid diseases: Personal or family history of medullary thyroid cancer, or uncontrolled hyperthyroidism/hypothyroidism 4.Gastrointestinal diseases: Having gastrointestinal surgery within 3 months, or inflammatory bowel disease or active gastric and duodenal ulcers 5.Pregnant or lactating women 6.Others: Type 1 diabetes, malignant tumors, severe cardiovascular diseases (such as NYHA IV).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
weight loss | 6 months